CLINICAL TRIAL: NCT06064708
Title: The Impact of Mindfulness-Based Intervention on Psychophysical Health in Patients Undergoing Hemodialysis: An Experimental Study
Brief Title: The Impact of Mindfulness-Based Intervention on Psychophysical Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jordan University of Science and Technology (Other)
Responsible Party: Principal Investigator, Hossam Najjem Alhawatmeh, Associate professor, Jordan University of Science and Technology
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 34/156/2023
Record Dates: First submitted 2023-09-26; First posted 2023-10-03 (Actual); Last update posted 2024-05-06 (Actual); Status verified 2024-05

CONDITIONS: End Stage Renal Disease
Keywords: Hemodialysis; Inflammatory Cytokines; Mindfulness-based intervention
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Intervention Model Description: the participants were randomly distributed into the experimental and control groups according to a straightforward 1:1 computer-generated sequence, giving them an equal chance of being in either of the two groups.
Who Masked: Investigator
Masking Description: A research assistant who did not participate in the other study phases collected the data, including blood sampling.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients with ESRD receiving mindfulness-based intervention (Experimental): Patients with ESRD who received mindfulness-based intervention: underwent hemodialysis thrice weekly, were at least 18 years old, were capable of reading and writing in Arabic, and agreed to participate. Patients under total parenteral nutrition (TPN), undergoing psychotherapy, taking psychopharmacological or anti-inflammatory drugs, and having immunocompromised and infectious illnesses were excluded from the research.
  Interventions: Behavioral: Mindfulness-based intervention
- Control group (No Intervention): The control group including patients with ESRD with the inclusion criteria similar to the experimental group received usual care, comprising biomedical normative dialysis treatment (the participants in this group did not receive any kind of additional treatment or holistic components). However, upon completion of the study, audio recordings of the intervention protocol were provided and explained to participants in the control group.

INTERVENTIONS:
Behavioral: Mindfulness-based intervention — The experimental group received 30 minutes of MBI according to Smith's (2005) MBI protocol, which is a standardized theory-based intervention.
  Smith's (2005) MBI protocol comprises six components:
  1. Being mindful of the breath (5 minutes).
  2. Being mindful of the body (5 minutes).
  3. Being mindful of the thought (5 minutes)
  4. Being mindful of the sound (5 minutes)
  5. Being mindful during walking (5 minutes)
  6. Full meditation (5 minutes).
  Arms: Patients with ESRD receiving mindfulness-based intervention

SUMMARY:
Background: Hemodialysis is considered as an effective therapy to remove harmful wastes from the body and to improve the quality of life in patients suffering from end-stage renal disease (ESRD). However, patients who receive hemodialysis perceive various stressors that are harmful to their physical and psychological well-being, particularly the immune system. Therefore, it is necessary to implement effective and practical therapeutic strategies to enhance the quality of life in this population. Mindfulness-based intervention is an effective mind-body connection program that is inadequately used in patients undergoing hemodialysis.

Objective: The current study aimed to investigate the effect of mindfulness-based intervention on physical and psychological symptoms (e.g., stress, anxiety, and depression) and pro-inflammatory biomarker levels (e.g., TNF, interleukin-6, and C-reactive protein) in patients with ESRD undergoing hemodialysis.

Method: Repeated measures, randomized, control experimental design was used. A convenience non-probability sampling technique to select the sample from the hemodialysis unit in the Princess Haya Bint AL_Hussine Hospital. The participants who were eligible and agreed to participate were randomly distributed into experimental (n = 31) and control (n = 30) groups. During their hemodialysis sessions, the experimental group' participants practiced 30-minute mindfulness-based intervention; three times a week for eight weeks). The Mindful Attention Awareness Scale (MAAS), Depression, Anxiety, and Stress Scale - 21 (DASS-21), Patient Health Questionnaire (PHQ-15), and serum blood levels (for tumor necrosis factor, interleukin-6, and C-reactive protein) were used to measure the dependent variables for both groups at baseline, after five weeks of the intervention, and at its end (eight weeks).

DETAILED DESCRIPTION:
Hemodialysis is considered as an effective and essential therapy to remove harmful wastes from the body and to improve the quality of life (QoL) of end-stage renal disease (ESRD) patients. However, patients undergoing hemodialysis experience multiple stressors (Finnegan-John & Thomas, 2013), negatively affecting their psychological and physical health, especially in relation to the immune system (Black & Slavich, 2016). Previous studies have indicated that patients undergoing maintenance hemodialysis experience a variety of physical and psychological symptoms (i.e., anxiety, fatigue, muscular spasms, and joint and bone pain), caused by a combination of stress, the disease itself, and intensive treatment (Hackett & Jardine, 2017; Hintistan, & Deniz, 2018), which has diverse effects including increased suicidal ideation (Yavuz, et al., 2022), impaired physical activity (Mallamaci et al., 2020), reduced QoL (Vasilopoulou et al., 2016), increased susceptibility to infectious disease (Maydych, 2019), and increased mortality and morbidity (Lv & Zhang, 2019).

High levels of blood proinflammatory markers, including C-reactive protein (CRP), tumor necrosis factor alpha (TNF-α), and interleukine-6 (IL-6), have been found in the majority of patients with ESRD (Abdel-Messeih et al., 2020; Park et al., 2022). The aetiology of inflammation in patients with ESRD is multidimensional, including patient-related causes, such as ESRD-related symptoms, comorbidity, and hemodialysis-related issues, especially those relating to the biocompatibility and quality of the dialysate and the dialysis membrane. These high levels of proinflammatory biomarkers in ESRDPs have been found to cause injury to other bodily organs in addition to the kidney, increasing morbidity and mortality (Abdel-Messeih et al., 2020).

Mind-body connection strategies such as mindfulness-based interventions (MBIs) are purposefully adopted in a wide range of structured interventions and have been proven to be highly effective in treating many physical and psychological symptoms of a wide range of psychiatric conditions associated with diverse chronic illnesses (Chu et al., 2021). MBIs reinforce adaptive coping processes and enhance positive reappraisal (Aliche & Onyishi, 2020). They enhance coping, reduce stress, improve mood and enhance the quality of spirituality and personal development in the adaptation of ESRD diagnosis and treatment (Sohn et al., 2018). They can also aid patients to be less reactive and to deal with fluctuating feelings through learning to accept the current experience more effectively, which ultimately reduces physical and emotional stress reactions (Chin-Lun Hung, 2019). Stress and emotional reactions are associated with increased levels of proinflammatory markers, whereby MBI could be effective in decreasing such markers by reducing stress and emotional reactions.

Many studies have demonstrated that MBI can improve psychophysical symptoms (i.e., stress, anxiety, depression, sleep disturbances, and pain) and pro-inflammatory markers (i.e., CRP, IL-6, and TNF α) in different psychiatric and medical populations (Aliche & Onyishi, 2020; Black & Slavich, 2016; Chu et al., 2021). A few studies have examined MBI's effects on limited numbers of psychophysical symptoms in ESRD patients undergoing hemodialysis, but they were hampered by severe limitations, such as small sample sizes and unstandardized intervention protocols.

For example, five weekly sessions of MBI improved perceived stress and QoL through the development of emotional regulation in patients undergoing hemodialysis (Alhawatmeh et al., 2022). Evidence has also shown that the practice of MBI reduced sleep disturbances, anxiety, stress, and depression in such patients (Alhawatmeh et al., 2022; Hackett & Jardine, 2017; Nejad et al., 2018). An extensive literature search did not find any previous study that examined the impact of MBI on serum proinflammatory biomarkers in patients with ESRD undergoing hemodialysis, although such interventions reduced proinflammatory markers such as CRP, interleukin-6 and TNF in different clinical conditions such as cancer, rheumatoid arthritis, and ulcerative colitis (Black & Slavich, 2016). Thus, the goal of this research is to investigate the effect of MBI on physical and psychological symptoms (e.g., stress, anxiety and depression) and proinflammatory biomarkers (e.g., TNF and CRP) in patients with ESRD undergoing hemodialysis.

Methodology

Design

A randomized, wait-list, control trial with two groups, and repeated measurement (RM) design was used in this randomized controlled trial (RCT).

Setting and Sample

The study was carried out in a military hospital located the Northern Jordan. It serves all patients, regardless of whether they have private, military, or public insurance. The hospital includes a dialysis unit with 30 dialysis machine beds and 112 patients are treated on average each week.

Convenience sampling initially recruited 64 participants, who were then randomly assigned by a researcher who was not involved in the patient assessment or recruitment process to the experimental (n=32) or control groups (n=32), using a simple 1:1 computer-generated sequence. However, 61 patients completed the study with 31 in the experimental group and 30 patients in the control group.

Determination of Sample Size

G*power 3.1.9.4 was used to calculate the sample size. Given a mixed-design repeated measures analysis of variance (ANOVA) (among groups and between groups), effect size of 0.25 and Cronbach's alpha coefficient of 0.05, and a power of 0.95, the recommended sample size is 44 patients. Taking into consideration a non-response and attrition rate of approximately 45%, as reported in a similar study (Alhawatmeh et al., 2022), the final required sample size was determined to be approximately 64 patients.

Procedure

After obtaining the IRB approval, the hospital managers were contacted by the study researcher to get approval for the study. After obtaining approval, the patients were contacted in person to describe the purpose of the study. Patients who decided to participate were asked to sign the consent form. After that, baseline measurements were taken in the hemodialysis unit in private contexts, where nobody else was present while participants filled out the questionnaire. A research assistant who did not participate in the other study phases collected the data, including blood sampling. This research assistant, who was an experienced registered nurse working in the hemodialysis unit for 10 years, followed strict infection control protocol during blood sampling.

After that, the participants were randomly distributed into the experimental and control groups according to a straightforward 1:1 computer-generated sequence, giving them an equal chance of being in either of the two groups. The foundation course was then conducted for the experimental group.

The MBI was delivered at the hospital, as described previously, and the participants in the experimental group were optionally advised to commit to practicing the study intervention program at home. Participants in both groups had to practice their normal routines of life before the study and not take psychiatric or alternative treatments to improve mood and notify the researcher if necessary.

Following baseline (Time 1), data was collected for the second and third time five and eight weeks after initiating the intervention (Time 2 and Time 3, respectively). All measurements were privately taken in similar situations and environments in the hemodialysis unit by the research assistant who took the baseline measurements. Nobody was present when participants filled out the questionnaire.

Data Analysis

SPSS version 25 was used to analyze the data. Descriptive statistics frequency, mean, and standard deviation were used as appropriate to describe the study participants. Repeated-measure ANOVA (RM ANOVA) (within-between-subject design) was used to test the study hypotheses. To assess whether there were significant mean differences between the study groups at each time measure and between the three-time measurements within each group, independent t-tests and repeated-measure ANOVA (between-subject only) respectively were conducted as post hoc testing.

Ethical Considerations

Jordan University of Science and Technology's Institutional Review Board (IRB) approved the proposed study. Participants who agreed to participate in the study were asked to sign a consent form that described the purpose and scope of the research. They confirmed that they had the freedom to reject participation in the study and that such rejection would not affect the care they received. They were assured that the research data would be stored in a secure location in a locked cabinet accessible only to the researcher, with numbers replacing their names to avoid their personal identification. No patients were excluded from the trial because of their gender, race, or nationality. During the intervention, if any patient felt dizzy or uncomfortable, the intervention was stopped, and the attending physician was informed immediately.

ELIGIBILITY:
Inclusion Criteria:

* Patients with ESRD who underwent hemodialysis thrice weekly
* were at least 18 years old
* were capable of reading and writing in Arabic
* agreed to participate.

Exclusion Criteria:

* Patients under total parenteral nutrition (TPN)
* undergoing psychotherapy
* taking psychopharmacological or anti-inflammatory drugs
* having immunocompromised and infectious illnesses

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2023-04-10 (Actual); Primary Completion 2023-08-10 (Actual); Study Completion 2023-08-30 (Actual)

PRIMARY OUTCOMES:
C-reactive protein | 8 weeks
  Serum CRP: This biomarker was analyzed using the ELISA protocol
Interleukin 6 | 8 weeks
  This biomarker was analyzed using the ELISA protocol
Tumor necrosis factor-alpha | 8 weeks
  This biomarker were analyzed using the ELISA protocol
Mindful Attention Awareness Scale (MAAS-15) | 8 weeks
  Mindful Attention Awareness Scale (MAAS-15) was used to assess dispositional mindfulness (Brown & Ryan, 2003). It includes 15 items measured on a six-point Likert-type scale, ranging from "almost always" (1) to "almost never" (6). The total score of the scale ranges from 15 to 90, with higher scores indicating a higher level of trait mindfulness. It is one-dimensional scale including 15 items measured on a six-point likert type scale, ranging from 1 (almost always) to 6 (almost never). The score range is between 15 and 90, with higher score indicting higher levels of mindfulness.
Depression, Anxiety and Stress Scale (DASS-21) | 8 weeks
  Depression, Anxiety and Stress Scale (DASS-21) was used to assess emotional symptoms (Antony et al., 1998). Each item is answered with a rating from 0 to 3, where 0 indicates "Did not apply to me", and 3 indicates "Applied to me most of the time". Total scores are calculated by summing the scores for the relevant items and then multiplying them by 2. The total scores for each subscale range from 0 to 42. Higher scores on the DASS-21 indicate a higher level of symptoms
Patient Health Questionnaire (PHQ-15) | 8 weeks
  Patient Health Questionnaire (PHQ-15) was used to measures the severity of 15 somatic symptoms (Kroenke et al., 2002). The PHQ-15 has a total score range of 0 to 30, whereby higher PHQ-15 scores are associated with more frequent and severe physical symptoms (Kroenke, et al., 2002)

CONTACTS AND LOCATIONS:
Locations (2):
- Jordan (2):
  - Hossam AlHawatmeh, Irbid, None Selected
  - Jordan University of Science and Technology, Irbid, None Selected

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Finnegan-John J, Thomas VJ. The psychosocial experience of patients with end-stage renal disease and its impact on quality of life: findings from a needs assessment to shape a service. ISRN Nephrol. 2012 Oct 21;2013:308986. doi: 10.5402/2013/308986. eCollection 2013. PMID 24959536
- [Background] Black DS, Slavich GM. Mindfulness meditation and the immune system: a systematic review of randomized controlled trials. Ann N Y Acad Sci. 2016 Jun;1373(1):13-24. doi: 10.1111/nyas.12998. Epub 2016 Jan 21. PMID 26799456
- [Background] Hackett ML, Jardine MJ. We Need to Talk about Depression and Dialysis: but What Questions Should We Ask, and Does Anyone Know the Answers? Clin J Am Soc Nephrol. 2017 Feb 7;12(2):222-224. doi: 10.2215/CJN.13031216. Epub 2017 Jan 26. No abstract available. PMID 28126705
- [Background] Hintistan, S., & Deniz, A. (2018). Cite this article as: Hintistan S, Deniz A. Evaluation of Symptoms in Patients Undergoing Hemodialysis. Bezmialem Science, 6, 112-120. https://doi.org/10.14235/bs.2018.1530
- [Background] Vasilopoulou C, Bourtsi E, Giaple S, Koutelekos I, Theofilou P, Polikandrioti M. The Impact of Anxiety and Depression on the Quality of Life of Hemodialysis Patients. Glob J Health Sci. 2015 May 17;8(1):45-55. doi: 10.5539/gjhs.v8n1p45. PMID 26234986
- [Background] Maydych V. The Interplay Between Stress, Inflammation, and Emotional Attention: Relevance for Depression. Front Neurosci. 2019 Apr 24;13:384. doi: 10.3389/fnins.2019.00384. eCollection 2019. PMID 31068783
- [Background] Abdel-Messeih PL, Alkady MM, Nosseir NM, Tawfik MS. Inflammatory markers in end-stage renal disease patients on haemodialysis. J Med Biochem. 2020 Oct 2;39(4):481-487. doi: 10.5937/jomb0-25120. PMID 33312065
- [Background] Chu SWF, Yeam CT, Low LL, Tay WY, Foo WYM, Seng JJB. The role of mind-body interventions in pre-dialysis chronic kidney disease and dialysis patients - A systematic review of literature. Complement Ther Med. 2021 Mar;57:102652. doi: 10.1016/j.ctim.2020.102652. Epub 2020 Dec 26. PMID 33373760
- [Background] Aliche JC, Onyishi IE. Mindfulness and wellbeing in older adults' survivors of herdsmen attack. The mediating effect of positive reappraisal. Aging Ment Health. 2020 Jul;24(7):1132-1140. doi: 10.1080/13607863.2019.1602592. Epub 2019 Apr 24. PMID 31016997
- [Background] Moosavi Nejad M, Shahgholian N, Samouei R. The effect of mindfulness program on general health of patients undergoing hemodialysis. J Educ Health Promot. 2018 Jun 12;7:74. doi: 10.4103/jehp.jehp_132_17. eCollection 2018. PMID 29963567
- [Background] Smith, J. (2005). Relaxation, meditation, & mindfulness: A mental health practitioner's guide to new and traditional approaches. https://books.google.com/books?hl=en&lr=&id=RCLr6ap7vRgC&oi=fnd&pg=PP11&dq=Smith,+J.+C.+(2005).+Relaxation,+meditation,+and+mindfulness:+A+mental+health+practitioner's+guide+to+new+and+traditional+approaches.+New+York,+NY,+Springer+Publishing+Co.&ots=vN4OeJpowy&sig=CZBq7fwjjxGVWb3139NndQtQ-xw
- [Background] Alhawatmeh H, Alshammari S, Rababah JA. Effects of mindfulness meditation on trait mindfulness, perceived stress, emotion regulation, and quality of life in hemodialysis patients: A randomized controlled trial. Int J Nurs Sci. 2022 Mar 8;9(2):139-146. doi: 10.1016/j.ijnss.2022.03.004. eCollection 2022 Apr. PMID 35509694
- [Background] Brown KW, Ryan RM. The benefits of being present: mindfulness and its role in psychological well-being. J Pers Soc Psychol. 2003 Apr;84(4):822-48. doi: 10.1037/0022-3514.84.4.822. PMID 12703651
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-15: validity of a new measure for evaluating the severity of somatic symptoms. Psychosom Med. 2002 Mar-Apr;64(2):258-66. doi: 10.1097/00006842-200203000-00008. PMID 11914441
- [Background] AlHadi AN, AlAteeq DA, Al-Sharif E, Bawazeer HM, Alanazi H, AlShomrani AT, Shuqdar RM, AlOwaybil R. An arabic translation, reliability, and validation of Patient Health Questionnaire in a Saudi sample. Ann Gen Psychiatry. 2017 Sep 6;16:32. doi: 10.1186/s12991-017-0155-1. eCollection 2017. PMID 28878812
- [Background] Igarashi NS, Karam CH, Afonso RF, Carneiro FD, Lacerda SS, Santos BF, Kozasa EH, Rangel EB. The effects of a short-term meditation-based mindfulness protocol in patients receiving hemodialysis. Psychol Health Med. 2022 Jul;27(6):1286-1295. doi: 10.1080/13548506.2021.1871769. Epub 2021 Jan 15. PMID 33449820
- [Background] Al-Dwaikat TN, Rababah JA, Al-Hammouri MM, Chlebowy DO. Social Support, Self-Efficacy, and Psychological Wellbeing of Adults with Type 2 Diabetes. West J Nurs Res. 2021 Apr;43(4):288-297. doi: 10.1177/0193945920921101. Epub 2020 May 16. PMID 32419665
- [Derived] Alhawatmeh H, Najadat I, Hweidi I, Abuhammad S. The impact of mindfulness meditation on pro-inflammatory biomarkers in patients with end-stage renal disease: A randomized trial. SAGE Open Med. 2024 Dec 18;12:20503121241308995. doi: 10.1177/20503121241308995. eCollection 2024. PMID 39713266
- [Derived] Alhawatmeh H, Najadat IA, Hweidi IM. Mindfulness-based intervention as a symptom management strategy in patients with end-stage renal disease: A controlled clinical trial. Int J Nurs Pract. 2024 Dec;30(6):e13282. doi: 10.1111/ijn.13282. Epub 2024 Jun 16. PMID 38880954